CLINICAL TRIAL: NCT03126409
Title: A Multicenter Randomized Trial to Compare the Graft Patency Between No-Touch Vein Harvesting Technique and Conventional Approach in Coronary Artery Bypass Graft Surgery: the PATENCY Study
Brief Title: No-Touch Versus Conventional Saphenous Vein Harvesting Technique
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20170414
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; coronary artery bypass graft
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-Touch vein harvesting technique (Experimental): During saphenous vein harvesting, surrounding tissue of the vein is preserved, and manual distension of the vein graft is avoided
  Interventions: Procedure: No-Touch vein harvesting technique
- Conventional vein harvesting (Active Comparator): During saphenous vein harvesting, surrounding tissue of the vein is stripped off, and manual distension is routinely performed
  Interventions: Procedure: Conventional vein harvesting

INTERVENTIONS:
Procedure: No-Touch vein harvesting technique — The No-Touch technique focuses on saphenous vein graft harvesting, featured by preserving the surrounding tissue of the vein while at the same time avoiding manual distension.
  Arms: No-Touch vein harvesting technique
Procedure: Conventional vein harvesting — During saphenous vein harvesting, surrounding tissue of the vein is stripped off, and manual distension is routinely performed
  Arms: Conventional vein harvesting

SUMMARY:
This study evaluates the short-term patency of vein graft harvested by the No-Touch technique compared to that by the conventional approach in patients undergoing isolated on-pump/off-pump coronary artery bypass graft (CABG) surgery. a total of at least 2000 patients undergoing isolated on-pump/off-pump CABG will be consecutively recruited from 7 hospitals across China and randomly assigned to receive No-Touch saphenous vein harvesting or conventional approach. All participants will be invited for clinical follow-up and 64-slice multislice computed tomography angiography (MSCTA) analysis at 3 months post-operatively.

DETAILED DESCRIPTION:
CABG is still the treatment of choice for ischemic heart disease. However, restenosis or occlusion may occur to graft vessels, leading to postoperative myocardial ischemia and subsequent clinical events. Long-term angiographic follow-up demonstrated that vein graft restenosis and occlusion are common among those receiving CABG, with a vein graft patency of less than 50% at 15 years postoperatively. Besides, it is found that graft occlusion may occur as early as 3 months after the surgery. It is, therefore, a major priority to improve the short-term postoperative vein graft patency so as to achieve better prognosis for patients.

Saphenous vein, the currently most frequently used graft material, occupies over 70% of all graft vessels.

Multiple factors may contribute to the early restenosis or occlusion of the vein grafts, including anastomosis technique, graft vessel quality, target lesion site and degree of stenosis, perioperative coagulating function, etc. The No-Touch technique focuses on saphenous vein graft harvesting, featured by preserving the surrounding tissue of the vein while at the same time avoiding manual distension. This technique has been reported associated with better short and long-term vein graft patency. However, these results mostly came from small-scale, single-center studies, therefore could hardly be recognized as high-level evidence for generalization of the technique.

This prospective multi-center study aims to compare the short-term saphenous vein graft patency harvested by the No-Touch technique and the conventional approach. This study will consecutively enroll 2000 patients undergoing isolated on-pump/off-pump CABG in 7 hospitals of China. After obtaining informed written consent, participants will be randomly allocated to either the No-Touch harvesting or conventional approach group. At baseline, participants will be interviewed to collect detailed information about on demographics, socioeconomic status, cardiovascular risk factors, clinical characteristics, treatments, in-hospital outcomes, general and disease-specific quality of life, function and mental status. During the follow-ups, the investigators will collect information about clinical outcomes events, long-term treatments, function, quality of life, symptoms, and medical care during the recovery period. All participants will be invited for 64-slice multi-slice computed tomography angiography (MSCTA) analysis at 3 months post-operatively for graft patency evaluation.

The patients, data adjudicators and CT reviewers will be blinded to the study. Due to the nature of this study, the operating surgeons, anesthetists and other operative room staff will not be blind in this study.

By comparing the short-term graft patency between the No-Touch and conventional vein harvesting groups, this study will contribute major evidence of the possible superiority of this technique, so as to improve patient outcomes after CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving first time isolated on-pump/off-pump CABG
* Patients with at least one available saphenous vein graft

Exclusion Criteria:

* Need for a concomitant cardiac or vascular surgeries (i.e. valve repair or replacement, Maze surgery)
* Redo-CABG
* Emergent CABG
* Using vascular stapler for anastomosis
* Endarterectomy of coronary artery during surgery
* Left ventricular repair due to ventricular aneurysm
* Combined with malignant tumor or other severe systemic conditions
* Severe renal insufficiency (i.e. creatinine >200 μmol/L)
* Contraindications for dual antiplatelet therapy, such as active gastroduodenal ulcer
* Participants of another ongoing clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2655 (Actual)
Dates: Start 2017-05-14 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of graft occlusion | 3 month after procedure
  All participants will be invited to return to their operating hospitals for 64-slice multi-slice computed tomography angiography to determine patencies of the graft vessels.

SECONDARY OUTCOMES:
Prevalence of graft occlusion | 1, 3, 5, 7, and 10 years after procedure
  All participants will be invited to return to their operating hospitals for 64-slice multi-slice computed tomography angiography to determine patencies of the graft vessels.
Overall major adverse cardiac or cerebrovascular events (MACCE) rate | 3 month , 1, 3, 5, 7, and 10 years after procedure
  MACCE includes death, myocardial infarction, stroke and/or repeat revascularization
Cardiac death | 3 month , 1, 3, 5, 7, and 10 years after procedure
  death from any heart disease
Documented non-lethal myocardial infarction | 3 month , 1, 3, 5, 7, and 10 years after procedure
  Myocardial infarction is defined according to the most recent guideline
Stroke | 3 month , 1, 3, 5, 7, and 10 years after procedure
  an acute symptomatic episode of focal or global neurological dysfunction caused by brain, spinal, or retinal vascular injury as a result of hemorrhage or infarction
Target lesion revascularization | 3 month , 1, 3, 5, 7, and 10 years after procedure
  CABG or percutaneous coronary intervention
Recurrence of Angina | 3 month, 1, 3, 5, 7, and 10 years after procedure
  recurrence of unstable angina
Rehospitalization due to cardiac reason | 3, 5, 7, and 10 years after procedure
  Rehospitalization due to cardiac reason

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academay of Medical Science and National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang X, Tian M, Zheng Z, Gao H, Wang Y, Wang L, Hu S. Rationale and design of a multicenter randomized trial to compare the graft patency between no-touch vein harvesting technique and conventional approach in coronary artery bypass graft surgery. Am Heart J. 2019 Apr;210:75-80. doi: 10.1016/j.ahj.2018.11.011. Epub 2018 Dec 6. PMID 30743210
- [Derived] Tian M, Wang X, Feng W, Wang H, Liu S, Liu Z, Chen Y, Miao Q, Su P, Li X, Wang Y, Lu B, Chen K, Zhang C, Hu S. No-touch versus conventional vein in coronary artery bypass grafting: three year follow-up of multicentre randomised PATENCY trial. BMJ. 2025 Apr 30;389:e082883. doi: 10.1136/bmj-2024-082883. PMID 40306935
- [Derived] Tian M, Wang X, Sun H, Feng W, Song Y, Lu F, Wang L, Wang Y, Xu B, Wang H, Liu S, Liu Z, Chen Y, Miao Q, Su P, Yang Y, Guo S, Lu B, Sun Z, Liu K, Zhang C, Wu Y, Xu H, Zhao W, Han C, Zhou X, Wang E, Huo X, Hu S. No-Touch Versus Conventional Vein Harvesting Techniques at 12 Months After Coronary Artery Bypass Grafting Surgery: Multicenter Randomized, Controlled Trial. Circulation. 2021 Oct 5;144(14):1120-1129. doi: 10.1161/CIRCULATIONAHA.121.055525. Epub 2021 Sep 13. PMID 34510911